CLINICAL TRIAL: NCT02523677
Title: Relationships Among Cognitive Function, Lifestyle, and Exercise After Cancer Treatment
Acronym: ReFLECT
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Edward McAuley, Shahid and Ann Carlson Khan Professor in Applied Health Sciences, University of Illinois at Urbana-Champaign
Other Study IDs: UIUC_IRB_15666
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Cognitive Impairment
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine relationships among lifestyle behaviors (i.e., physical activity, sleep), cognitive function (i.e., memory, processing speed, and executive function), and quality of life in breast cancer patients and survivors across time. The investigators will compare the strength of these relationships across age cohorts and time since treatment and diagnosis. Participants will complete a battery of questionnaires and a set of cognitive tests on an iPad app specifically tailored for this study. A subset of participants will also wear an accelerometer for seven days. Data will be collected at baseline and 6-month follow-up.

This research is critical to identifying potentially important approaches to improving health outcomes and quality of life in breast cancer patients and survivors. Previous research provides evidence of the influence of lifestyle behaviors on cognition and quality of life in healthy aging populations. However, despite data indicating cancer's negative impact on lifestyle behaviors, cognition, and quality of life, very few studies have investigated interactions among these factors in cancer patients and survivors.

DETAILED DESCRIPTION:
Interested individuals will visit the ReFLECT Study website (www.reflectstudies.org) to learn more about the study and receive instructions on how to participate. Individuals will be instructed to create a username (email address) and password for BrainBaseline© (www.BrainBaseline.com; Digital Artefacts, Iowa City, IA). While BrainBaseline© is a commercially available mobile app, a version specifically tailored for this study will be used. The website directions will include information on how to download the BrainBaseline© iPad app (for ReFLECT) from the iTunes store. Each time a participant closes and reopens the iPad app, she will be required to enter her BrainBaseline© username and password. Upon opening the iPad app for the first time, the individual will be asked to confirm their eligibility for the study. If eligible, the individual will proceed to the consent form. Participants will electronically sign the Institutional Review Board-approved informed consent form before completing a battery of questionnaires assessing demographics, medical history, physical activity, sedentary behavior, sleep, fatigue, quality of life, satisfaction with life, depressive symptoms, and perceived memory. Individuals cannot view the questionnaires until they have electronically signed the consent form. Participants will also be asked to complete a set of ten evidence-based cognitive tests assessing attention, speed of processing, and executive function. Descriptions of the tests are available at www.BrainBaseline.com/assessments. The questionnaires are expected to take approximately 45 minutes and the cognitive tests are expected to take approximately 60 minutes to complete. Participants will be instructed to complete the questionnaires and cognitive tests within two weeks of signing the consent form. The onscreen instructions and consent form will also notify participants that a) they do not have to complete either the questionnaires or the cognitive tests in one sitting, but can return to them during the course of the week, and b) they can move back and forth between the questionnaires and cognitive tests (i.e., do not need to finish one section before moving to the next). Reminder emails will be sent on days 7 and 10 to remind participants to complete assessments.

A subset of participants who volunteer to do so will also wear an accelerometer for 24 hours per day for 7 consecutive days to objectively measure activity levels and sleep quality. Individuals will be asked if they are willing to be contacted to wear the accelerometer via the consent form. Only those individuals who check the box agreeing to be contacted by the research team will be contacted to wear the accelerometer (see consent form). Participants will be contacted via email and instructed to reply to the researcher by phone or email with their mailing address. The accelerometer, instructions for wear, a Record of Use form, and a postage-paid return envelope will be mailed to participants who agree to wear the monitor. Mailing labels from postage-paid return envelopes will be disposed of after accelerometers have been returned and recorded. The accelerometer will be worn during women's daily life on a normal week; therefore, minimal additional time committed to research activities will be required of participants. No contact will be solicited with participants over the course of the 6-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Female diagnosed with breast cancer
* 21 years or older
* English speaking
* Access to an iPad with iOS 6.2 or later and the Internet

Exclusion Criteria:

* Male
* Individuals under 21 years of age
* Individuals who do not have access to an iPad with iOS 6.2 or later

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients and survivors aged 21 years or older and who have access to an iPad and the Internet.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Executive Function | Baseline, 6 months
  Executive Function will be expressed as a composite score of the following cognitive tests: Flanker, Task-Switch, Trails A&B, Mazes
Change in Working Memory | Baseline, 6 months
  Working Memory will be expressed as a composite score of the following cognitive tests: N-Back, Spatial Working Memory, Spatial Span, and Swap
Change in Speed of Processing | Baseline, 6 months
  Speed of Processing will be expressed as a composite score of the following cognitive tests: Digital Symbols Substitution, Flanker, Speed, Task-Switch, and Trails A&B

SECONDARY OUTCOMES:
Medical Health History | Baseline, 6 months
  Medical health history will be measured at baseline and 6-month follow-up to identify any changes to participants' health status during the study period. If no changes are observed, baseline values may be used as covariates or moderators in data analyses.
Change in Sleep Quality (objectively measured) | Baseline, 6 months
  Change in sleep quality as measured by a wrist-worn accelerometer will be examined as a predictor of change in executive function, working memory, and speed of processing.
Change in Physical Activity (objectively measured) | Baseline, 6 months
  Change in physical activity as measured by a waist-worn accelerometer will be examined as a predictor of change in executive function, working memory, and speed of processing.

OTHER OUTCOMES:
Change in Sleep Quality (self-report) | Baseline, 6 months
  Change in sleep quality as measured by the Pittsburgh Sleep Quality Index will be examined as a predictor of change in executive function, working memory, and speed of processing.
Change in Physical Activity (self-report) | Baseline, 6 months
  Change in physical activity as measured by the Godin Leisure-Time Exercise Questionnaire will be examined as a predictor of change in executive function, working memory, and speed of processing.
Change in Sitting Time | Baseline, 6 months
  Change in sitting time as measured by the Sitting Time Questionnaire will be examined as a predictor of change in executive function, working memory, and speed of processing.
Change in Sedentary Activity | Baseline, 6 months
  Change in sedentary activity as measured by the Longitudinal Aging Study Amsterdam Sedentary Behavior Questionnaire will be examined as a predictor of change in executive function, working memory, and speed of processing.
Change in Current Symptoms | Baseline, 6 months
  Change in breast cancer related symptoms as measured by the Functional Assessment of Cancer Therapy - Breast will be examined as a potential confounder or moderator of the relationship between physical activity and cognitive function.
Change in Fatigue | Baseline, 6 months
  Change in fatigue as measured by the Functional Assessment of Chronic Illness Therapy 13-Item Fatigue Scale will be examined as a potential confounder or moderator of the relationship between physical activity and cognitive function.
Change in Anxiety and Depression | Baseline, 6 months
  Change in anxiety and depression as measured by the Hospital Anxiety and Depression Scale will be examined as potential confounders or moderators of the relationship between physical activity and cognitive function.
Change in Quality of Life | Baseline, 6 months
  Relationships between change in physical activity and cognitive function and change in quality of life as measured by the Satisfaction with Life Scale will be examined.
Change in Memory | Baseline, 6 months
  Change in memory as measured by the Memory Controllability Inventory will be examined as an outcome of changes in sleep quality and physical activity.
Change in Forgetfulness | Baseline, 6 months
  Change in forgetfulness as measured by the Frequency of Forgetting Questionnaire will be examined as an outcome of changes in sleep quality and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Marshall AL, Miller YD, Burton NW, Brown WJ. Measuring total and domain-specific sitting: a study of reliability and validity. Med Sci Sports Exerc. 2010 Jun;42(6):1094-102. doi: 10.1249/MSS.0b013e3181c5ec18. PMID 19997030
- [Background] Visser M, Koster A. Development of a questionnaire to assess sedentary time in older persons--a comparative study using accelerometry. BMC Geriatr. 2013 Jul 30;13:80. doi: 10.1186/1471-2318-13-80. PMID 23899190
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Lachman ME, Bandura M, Weaver SL, Elliott E. Assessing memory control beliefs: The Memory Controllability Inventory. Aging Cogn 2(1):67-84, 1995.
- [Background] Zelinski EM, Gilewski MJ. A 10-item Rasch modeled memory self-efficacy scale. Aging Ment Health. 2004 Jul;8(4):293-306. doi: 10.1080/13607860410001709665. PMID 15370046
- [Background] Eriksen BA, Eriksen CW. Effects of noise letters upon identification of a target letter in a non-search task. Perception and Psychophysics. 16:143-149, 1974.
- [Background] Awh E, Jonides J, Reuter-Lorenz PA. Rehearsal in spatial working memory. J Exp Psychol Hum Percept Perform. 1998 Jun;24(3):780-90. doi: 10.1037//0096-1523.24.3.780. PMID 9627416
- [Background] KIRCHNER WK. Age differences in short-term retention of rapidly changing information. J Exp Psychol. 1958 Apr;55(4):352-8. doi: 10.1037/h0043688. No abstract available. PMID 13539317
- [Background] Basner M, Dinges DF. Maximizing sensitivity of the psychomotor vigilance test (PVT) to sleep loss. Sleep. 2011 May 1;34(5):581-91. doi: 10.1093/sleep/34.5.581. PMID 21532951
- [Background] Monsell S. Task switching. Trends Cogn Sci. 2003 Mar;7(3):134-140. doi: 10.1016/s1364-6613(03)00028-7. PMID 12639695
- [Derived] Ehlers DK, Fanning J, Sunderlage A, Severson J, Kramer AF, McAuley E. Influence of sitting behaviors on sleep disturbance and memory impairment in breast cancer survivors. Cancer Med. 2020 May;9(10):3417-3424. doi: 10.1002/cam4.3008. Epub 2020 Mar 23. PMID 32202706
- [Derived] Ehlers DK, Fanning J, Salerno EA, Aguinaga S, Cosman J, Severson J, Kramer AF, McAuley E. Replacing sedentary time with physical activity or sleep: effects on cancer-related cognitive impairment in breast cancer survivors. BMC Cancer. 2018 Jun 25;18(1):685. doi: 10.1186/s12885-018-4603-3. PMID 29940894